CLINICAL TRIAL: NCT01522885
Title: KatGuide-trial. KatGuide Method Versus Conventional Method at Insertion of Chest Tube. A Randomized, Parallel Group, Controlled Trial.
Brief Title: KatGuide Method Versus Conventional Method at Insertion of Chest Tube
Acronym: KatGuide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Niels Katballe (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Niels Katballe, Coordinating investigator, MD, PhD, University of Aarhus
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011375
Record Dates: First submitted 2012-01-24; First posted 2012-02-01 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Pneumothorax; Hydrothorax; Hemothorax; Empyema; Chylothorax
Keywords: Chest tube; placement; mal positioning
MeSH Terms: conditions — Pneumothorax; Hydrothorax; Hemothorax; Empyema; Chylothorax | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KatGuide (Active Comparator): Chest tube insertion is performed by using the KatGuide
  Interventions: Device: KatGuide versus conventional method (forceps)
- Conventional group (Active Comparator): Chest tubes are inserted by using conventional method (forceps) for large bore chest tube insertion.
  Interventions: Procedure: Chest tube insertion

INTERVENTIONS:
Device: KatGuide versus conventional method (forceps) — According to randomization Chest tubes are placed in the pleural cavity by using the KatGuide device.
  Arms: KatGuide
Procedure: Chest tube insertion — The chest tube is placed in the pleural cavity by using a forceps (conventional method) or KatGuide
  Arms: Conventional group

SUMMARY:
The purpose of this study is to investigate whether if KatGuide (a new developed medical device) improves the placing of a large bore chest tube in the pleural cavity compared to the conventional method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pneumothorax in the upper pleural space or fluid in the lower pleural space.
* Indication for upper or lower placement of a single chest tube in the pleural cavity
* 18 years of age or older

Exclusion Criteria:

* Fertile women
* Patients who can not give written or verbal consent to participate
* If there is no time or possibility to inform the patient
* Patients who already has a large bore chest tube
* Patients with long lasting (>14 days) or chronic chest tube
* Patients with both fluid and air in the pleural cavity
* Patients where "the safe area" (front axillary fold, IC 4-5) can not be used for chest tube insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Chest tube placement | 3 hours
  X-ray examination of the chest is performed within 3 hours after the chest tube insertion, to evaluate if the placement of the chest tube is acceptable.

SECONDARY OUTCOMES:
Length of hospital stay | 5 days
  The hospital stay depends on how long time it takes to solve the chest tube related problem. In a few patients it takes only one day, but in severe cases it may take weeks before the patient can be discharged. We predict, that the patient will be in hospital for a mean time of 5 days.
Time with chest tube | 3 days (mean time)
  A few patients can have the chest tube removed in only one day, but some patients must have a chest tube for weeks. We predict that the patients will have a chest tube in a mean time of 3 days.
Infection in wound | 4 weeks
  4 weeks after the chest tube insertion, the patient is contacted and the patient is asked whether there are problems with infection of the wound.
Number of chest tubes | 7 days (mean time)
  It is observed whether the patient has multiple chest tubes inserted in the pleural cavity at the same side. It is predicted, that these patients are hospitalized longer than patients with only one chest tube. We predict, that these patients are hospitalized for a mean time of 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Katballe, MD, PhD, Study Director — University of Aarhus
Locations (4):
- Denmark (4):
  - Niels Katballe, Aarhus, Aarhus N
  - Vytautas Nekrasas, Aalborg, Denmark
  - Niels Katballe, Aarhus N, Denmark
  - Peter B Licht, Odense, Denmark

REFERENCES:
- [Derived] Katballe N, Moeller LB, Olesen WH, Litzer MM, Andersen G, Nekrasas V, Licht PB, Bach P, Pilegaard HK. A Novel Device for Accurate Chest Tube Insertion: A Randomized Controlled Trial. Ann Thorac Surg. 2016 Feb;101(2):527-32. doi: 10.1016/j.athoracsur.2015.07.017. Epub 2015 Sep 26. PMID 26409714